CLINICAL TRIAL: NCT00001122
Title: A Phase II, Randomized, Open-Label Study of Maximally Assisted Therapy (MAT) Compared to Self-Administered Therapy (SAT) for the Treatment of HIV Infection in Antiretroviral Naive Subjects With CD4 Greater Than or Equal to 200 Cells/mm3
Brief Title: A Study of an Adherence Plan to Help HIV-Positive Patients Take Their First Anti-HIV Medications Correctly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Crossover | Purpose: Treatment
Other Study IDs: AIEDRP AI-05-003; AEHIV 003: MAT
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2005-01

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Nelfinavir; Reverse Transcriptase Inhibitors; Self Care; Anti-HIV Agents; Viral Load; efavirenz; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; efavirenz; Stavudine; Didanosine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if observed therapy can help HIV-positive patients stick to their anti-HIV medication schedule. Observed therapy means that a nurse will watch patients take their medications to make sure that they take them correctly.

It is very important that HIV-positive patients take their anti-HIV medications correctly so they get the best possible benefit from them. Taking the drugs correctly, called "adherence," may keep HIV virus levels in the blood (viral load) low for a longer time. Adherence can also slow the development of drug resistance, and this is especially important in patients with early HIV infection who are just beginning treatment. However, anti-HIV medication schedules are often complicated, and many patients have difficulty remembering to take their drugs at the correct time. This study will look at the effectiveness of a plan to help patients with this problem.

DETAILED DESCRIPTION:
Novel approaches are needed to improve adherence to combination antiretroviral therapy. Nonadherence can lead to reduced drug levels and inadequate viral suppression, which accelerates drug resistance. Thus nonadherence in the first few months of primary HIV infection can limit therapeutic options for an individual years later. Barriers to optimal treatment adherence in patients with early HIV infection include complex treatment regimens which disrupt daily routines, drug intolerance, and concomitant illness including depression. Directly observed therapy has been successful in improving overall effectiveness of antituberculosis therapy and may be a useful strategy in HIV-infected patients.

All patients receive combination antiretroviral therapy with didanosine (ddI), stavudine (d4T), efavirenz (EFV), and nelfinavir (NFV). Patients are randomized to self-administered (SAT) versus observed (MAT) therapy for 24 weeks. Patients randomized to MAT receive one directly observed dose (ddI, d4T, EFV, and NFV) of their antiretroviral regimen by a field worker or nurse at the clinic 5 days per week. As a reminder for the second NFV and d4T dose, MAT patients are provided with an alarm watch programmed to sound at dosing times. The alarm watch also serves as a reminder for weekend doses that will not be directly observed. Patients randomized to SAT receive standard care. All patients are monitored with monthly plasma HIV RNA levels and CD4 and CD8 cell counts. At Week 24, all patients are crossed over to SAT for an additional 48 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 13 years old (consent is required if you are under 18).
* Have a CD4 count of at least 200 cells/mm3 within 30 days of study entry.
* Have never taken anti-HIV drugs.
* Agree to practice effective methods of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have cancer (except for Kaposi's sarcoma) that requires treatment.
* Have a history of hepatitis or pancreatitis.
* Have peripheral neuropathy.
* Have an alcohol abuse problem.
* Are pregnant or breast-feeding.
* Are taking certain medications, such as rifabutin, rifampin, interleukin, or chemotherapy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74
Dates: Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Little, Principal Investigator; Diane Havlir, Principal Investigator
Locations (2):
- United States (2):
  - UCSD, San Diego, California
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas